CLINICAL TRIAL: NCT03509025
Title: Open, Multicenter Follow-up Trial About Active Group of Phase IIb Clinical Trial of JOINTSTEM in Patients With Degenerative Arthritis
Brief Title: Follow-up Study for Participants Jointstem Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JM2b-FU
Record Dates: First submitted 2017-03-13; First posted 2018-04-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long Term Follow-up after Jointstem Transplantation (Experimental)
  Interventions: Drug: Jointstem

INTERVENTIONS:
Drug: Jointstem — JOINTSTEM is an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is incubated without additional genetic modification or mechanical and chemical modification through differentiation, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.
  Other Names: autologous adipose-derived mesenchymal stem cells

SUMMARY:
This study is a long term follow-up study to investigate the safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with Knee Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent in writing to participate in the study by signing and dating an informed consent document
* Patients who transplanted Jointstem on phase 2b clinical trial

Exclusion Criteria:

* Preparing for Pregnancy or Pregnant women or lactating mothers.
* Patients who the principal investigator considers inappropriate for the clinical tria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 60 months
  Incidence of adverse events from baseline to 60 months

SECONDARY OUTCOMES:
WOMAC score | Baseline and 12 months
  Change from baseline on WOMAC (Western Ontario and McMaster Universities Arthritis Index) score
WOMAC 3 subscale score | Baseline and 12 months
  Change from baseline on WOMAC 3 subscale (Pain, stiffness, and physical function) score
X-ray | Baseline and 12 months
  X-ray perform to measure with Kellgren-Lawrence grade

CONTACTS AND LOCATIONS:
Overall Officials: KangIl Kim, M.D., Ph.D., Principal Investigator — KyungHee University Gangdong Hospital
Locations (2):
- South Korea (2):
  - KyungHee University Gangdong Hospital, Seoul
  - GangNam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No